CLINICAL TRIAL: NCT05098977
Title: The Usefulness of Assessing Heart Rate Variability in Patients With Acute Myocardial Infarction: From Primary Angioplasty to Secondary Long-term Prevention - a Single Centre, Prospective, Observational Cohort Study
Brief Title: The Usefulness of Assessing Heart Rate Variability in Patients With Acute Myocardial Infarction
Acronym: HeaRt-V-AMI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Grigore T. Popa University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Professor Adrian Covic, Professor coordinator, Grigore T. Popa University of Medicine and Pharmacy
Other Study IDs: HeaRt-V-AMI
Record Dates: First submitted 2021-10-18; First posted 2021-10-29 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Myocardial Infarction; Autonomic Dysfunction
Keywords: Heart rate variability; Percutaneous coronary intervention; Drug-eluting stents; Risk assessment; Prognosis; Major adverse cardiovascular events; Left ventricular ejection fraction; Secondary prevention
MeSH Terms: conditions — Myocardial Infarction; Primary Dysautonomias | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — CK-MB, AST, LDH, cardiac-specific troponin, glycemia, glycosylated hemoglobin, lipid profile, complete blood count, hemoglobin, hematocrit, serum urea and creatinine (estimated glomerular filtration rate using CKD-EPI equation), serum potassium and sodium, sideremia, plasma ferritin, thyroid-stimulating hormone, serum thyroxine, C-reactive protein, N-terminal pro b-type natriuretic peptide.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Heart rate variability measurement — HRV will be measured at the moment of patients' admission to the cardiac catheterization laboratory on the top of therapy guided by European guidelines. Both, time- and frequency-domain parameters (respectively, SDNN, SDANN, RMSSD and LF, HF, LF/HF ratio) of the HRV will be obtained using a validated medical device during 5-minute segments before and after revascularization of the culprit artery. In addition, HRV will be evaluated in ambulatory setting, at 1 month and at 6 months after the index event. Obtained interbeat interval data will be further analysed using a dedicated software in order to derive specified HRV parameters.
Procedure: Percutaneous coronary intervention — Coronary angiography and PCI will be performed using femoral or radial approach after local anesthetic infiltration with Lidocaine and arterial sheath placement. Following the culprit lesion detection and guidewire placement, thromboaspiration and glycoprotein IIb/IIIa inhibitors will be left to the operator decision. Also, the choice of coronary stenting technique and stent sizing will be performed according to the operator experience. Antiplatelet and anticoagulant drugs will be administered in concordance with latest European guidelines.
  Other Names: PCI

SUMMARY:
Aims

* heart rate variability (HRV) assessment in patients with acute myocardial infarction who undergo primary percutaneous coronary intervention (PCI);
* measurement of HRV using a device approved for medical use in Europe;
* assessment of the correlation between HRV and short- and long-term adverse cardiovascular events (composite of all-cause mortality and major adverse cardiovascular events - MACE; ventricular arrhythmias; hospital admissions for heart failure; left ventricular systolic and diastolic disfunction; MACE in special subgroups of patients - elderly, diabetes mellitus, chronic kidney disease) in patients treated by primary PCI for acute myocardial infarction;
* creating a registry of HRV parameters measured in a contemporary cohort of patients with acute myocardial infarction.

DETAILED DESCRIPTION:
The following data will be collected:

* general demographic data;
* time from chest pain onset to primary PCI;
* comorbidities (ischemic heart disease, arterial hypertension, previous PCI or coronary artery bypass surgery - CABG, heart failure, peripheral artery disease, atrial fibrillation, stroke, diabetes mellitus, kidney disease);
* cardiovascular risk factors (age, body mass index, smoking, abdominal perimeter, sedentarism, gender, inflammation);
* cardiac rhythm derived from electrocardiographic data;
* HRV time- and frequency domain parameters (respectively, SDNN, SDANN, RMSSD and LF, HF, LF/HF ratio);
* routine biological data and biomarkers, including creatine kinase-MB (CK-MB), aspartate transaminase (AST), lactate dehydrogenase (LDH) and cardiac-specific troponin;
* left ventricular ejection fraction at admission, at discharge and at follow-up (1 month, 6 months and 1 year);
* initial and final thrombolysis in myocardial infarction (TIMI) flow;
* type of stent used for coronary angioplasty;
* Global Registry of Acute Coronary Events (GRACE) score;
* SYNTAX score II in case of three-vessel coronary disease or involving left main stem;
* in-hospital, one month and long-term clinical outcomes (composite of all-cause mortality and major adverse cardiovascular events - MACE; ventricular arrhythmias; hospital admissions for heart failure; left ventricular systolic and diastolic disfunction; MACE in special subgroups of patients - elderly, diabetes mellitus, chronic kidney disease).

ELIGIBILITY:
Inclusion Criteria:

* patients with ST-Elevation Myocardial Infarction (STEMI) treated with primary PCI within 12 hours from symptoms onset;
* patients in sinus rhythm;
* patients who have read and signed the standard informed consent regarding enrolment in the study.

Exclusion Criteria:

* unconscious or intubated patients who are unable to sign the standard informed consent;
* patients with atrial fibrillation;
* patients with sinus node dysfunction or atrioventricular block of any degree;
* frequent premature supraventricular or ventricular contractions;
* paced ventricular rhythm;
* patients treated with positive inotropic and chronotropic drugs;
* history of myocardial infarction or myocardial revascularization (PCI or CABG);
* patients refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with STEMI referred to catheterization laboratory from Institute of Cardiovascular Diseases "Prof. George IM Georgescu", Iasi, within 12 hours from symptoms onset.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Composite of all-cause mortality and major adverse cardiovascular events (MACE) | in-hospital, 1 month and 1 year
  MACE will be defined as cardiac mortality, fatal and non-fatal myocardial infarction, unplanned target vessel revascularization and stroke)

SECONDARY OUTCOMES:
All-cause mortality | in-hospital, 1 month and 1 year
  Defined as total number of deaths from any cause
Cardiac mortality | in-hospital, 1 month and 1 year
  Defined as number of deaths due to cardiac causes
Fatal and non-fatal myocardial infarction | in-hospital, 1 month and 1 year
  Defined as a new myocardial infarction
Target vessel revascularization | in-hospital, 1 month and 1 year
  Defined as unplanned PCI or coronary artery bypass graft surgery for a stenosis in another part of the vessel treated at the index PCI
Target lesion revascularization | in-hospital, 1 month and 1 year
  Defined as repeat PCI or coronary artery bypass graft surgery of the target lesion treated at the index PCI
Stroke | in-hospital, 1 month and 1 year
  Defined as ischemic or hemorrhagic stroke

OTHER OUTCOMES:
Hospital admissions for heart failure | 1 year
  Defined as any subsequent admission for a primary diagnosis of heart failure
Ventricular arrhythmias | in-hospital, 1 month and 1 year
  Defined as electrocardiographic documentation of ventricular fibrillation or sustained ventricular tachycardia
Left ventricular ejection fraction (LVEF) | in-hospital, 1 month and 1 year
  Appraised using two-dimensional transthoracic echocardiography - Simpsons method
Left ventricular diastolic dysfunction | in-hospital, 1 month and 1 year
  Appraised using two-dimensional transthoracic echocardiography - E/A and E/e prime ratios
Composite of all-cause mortality and major adverse cardiovascular events in special subgroup of patients | in-hospital, 1 month and 1 year
  elderly, diabetes mellitus, chronic kidney disease

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Covic, Professor, Study Chair — Gr T Popa University of Medicine and Pharmacy Iasi ROMANIA
Locations (1):
- Department of Interventional Cardiology, Institute of Cardiovascular Diseases "Prof. George IM Georgescu" Iasi, Iași, Romania